CLINICAL TRIAL: NCT06972940
Title: A Prospective, Multicenter, Randomized, No-treatment Controlled, Assessor-blinded, Superiority Clinical Trial to Evaluate the Efficacy and Safety of Polycaprolactone Gel for Injection to Improve Temple Hollowing in Chinese Adults
Acronym: Ellanse M
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AQTIS Medical B.V. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HDM6007; HDM6007 (Other Grant/Funding Number: Sinclair Pharmaceuticals (Hangzhou) Co., Ltd.)
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Temple Hollowing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the method of endpoint blind evaluation is adopted, that is, it's blinded for the evaluator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Polycaprolactone (PCL) Based Facial Injectable (Experimental): Experimental: Polycaprolactone (PCL) Based Facial Injectable
  Interventions: Device: Polycaprolactone (PCL) Based Facial Injectable
- No treatment control (No Intervention): No treatment control

INTERVENTIONS:
Device: Polycaprolactone (PCL) Based Facial Injectable — Polycaprolactone (PCL) Based Facial Injectable
  Arms: Experimental: Polycaprolactone (PCL) Based Facial Injectable

SUMMARY:
A Prospective, Multicenter, Randomized, No-treatment controlled, Assessor-blinded, Superiority Clinical Trial to Evaluate the Efficacy and Safety of Polycaprolactone Gel for Injection to Improve Temple Hollowing in Chinese Adults

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 65 years old (inclusive), male or female;
2. Subjects who are willing to receive temple filling treatment;
3. Subjects with flat to severe temple hollowing on both sides (i.e. ATHS scores of 1- 4 on two sides, which are not necessarily the same but should have a difference of at most 2) as assessed by the blinded investigators;
4. Subjects able to self-assess efficacy without spectacles or with contact lenses;
5. Subjects who voluntarily sign the ICF, understand and accept the duration of the study, and will be able and willing to comply with all requirements, including scheduled treatment, follow-up, and other study procedures

Exclusion Criteria:

1. With known allergic reactions to polycaprolactone (PCL),carboxymethylcellulose (CMC), glycerin or any ingredient in the product;
2. With known history of severe allergic reactions and multiple severe allergies;
3. With abnormal coagulation mechanism (activated partial thromboplastin time (APTT) > 1.5 times the upper limit of normal) at screening, or having received any thrombolytic agent, anticoagulant, or antiplatelet drug (e.g.,warfarin, aspirin) within 2 weeks prior to enrollment;
4. With temple hollowing due to trauma, congenital malformation, or congenital or acquired lipodystrophy;
5. With previous or current temporal arteritis;
6. With temporomandibular disorders or other mandibular diseases;
7. With recurrent temporal headaches, such as temporal tendonitis, and migraine;
8. Having received injection of polymethyl methacrylate, silicone, expanded polytetrafluoroethylene, autologous fat, or any other fillers in the temple;
9. Having received injection of calcium hydroxyapatite, poly-L-lactic acid, polycaprolactone, or any other fillers in the temple within 2 years before enrollment;
10. Having received injection of crosslinked HA or any other unknown materials above the subnasale within 12 months before enrollment (except the injections in nasolabial folds and mid-face);
11. Having received collagen injection above the subnasale within 6 months before enrollment (except the injections in nasolabial folds and mid-face);
12. Having received injection of non-crosslinked sodium hyaluronate (including skin boosters), short wave therapy, ultrasound therapy, laser or chemical peeling, dermabrasion, or any other treatment within 3 months before enrollment;
13. Having received face lifting (thread lift) above the subnasale within 12 months before enrollment;
14. Having received radio frequency therapy or botulinum toxin injection above the subnasale within 6 months before enrollment, such as periorbital rhytidectomy, and treatment of masseteric hypertrophy (except the injections in nasolabial folds and mid-face) ;
15. Having ever received surgery in the temples, which affects efficacy evaluation as judged by the investigator;
16. Having tattoos, piercings, significant facial hair (e.g., whiskers), scars, deformities, unhealed wounds, active skin diseases or inflammation or infections (e.g., herpes, acne, eczema, dermatitis, psoriasis, and herpes zoster), abscess, cancers or precancerous lesions, etc. above the subnasale that may affect the efficacy evaluation or increase treatment-related risk;
17. Subjects with active autoimmune diseases or medical history (e.g. systemic lupus erythematosus, rheumatoid arthritis, scleroderma, dermatomyositis, etc.), active sepsis, and porphyria;
18. Subjects with a tendency to form keloids, hypertrophic scars, or any other healing disorders;
19. Having received chemotherapy, immunosuppressants, immunomodulatory therapy (e.g., monoclonal antibodies) or systemic corticosteroids (except inhaled corticosteroids) within 3 months prior to enrollment;
20. Subjects with severe dysfunction of vital organs (brain, heart, lung, liver, kidney, etc.), such as serious cardiovascular and cerebrovascular diseases, serious lung diseases, liver function (ALT, AST) > 2 times ULN, renal function (Cr) > 1.5 times ULN, uncontrolled diabetes mellitus or epilepsy, and other conditions, as judged by the investigator;
21. Subjects who plan to receive filling, wrinkle correction, or surgery at any site above the subnasale during the study period;
22. Subjects who received orthodontics, dental implants, denture installation, and any other operations or surgical treatments that affect the upper facial contour within 1 year before enrollment, or are receiving such operations or surgical treatments, or plan to receive such operations or surgical treatments during the study period;
23. Subjects who plan to have an obvious weight change (≥10%) within the study period;
24. Having participated in other clinical trials within 3 months prior to enrollment in this study or being currently participating in other clinical trials;
25. Pregnant or lactating women;
26. Women of childbearing potential who plan to become pregnant or fail to use effective contraceptive measures during the study** (female subjects ofchildbearing potential should have a negative pregnancy test prior to the first injection) and male subjects who plan to have a child or are unwilling to use appropriate contraceptive measures;
27. Those who are inappropriate to participate in this clinical study in the opinion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-10-12 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint: Response rate of temple hollowing improvement at Month 12 (Month 12 after the last injection in the test group and Month 12 after randomization in the control group, as assessed by a blinded investigator) | Primary efficacy endpoint: Response rate of temple hollowing improvement at Month 12 (Month 12 after the last injection in the test group and Month 12 after randomization in the control group, as assessed by a blinded investigator)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No